CLINICAL TRIAL: NCT03824041
Title: Aronia Berry Supplementation for Improving Vascular Endothelial Dysfunction and Modulating the Gut Microbiota in Middle-Aged/Older Adults
Brief Title: Effects of Aronia Berries on Vascular Endothelial Function and the Gut Microbiota in Middle-Aged/Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Naturex-Dbs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-8045H
Record Dates: First submitted 2019-01-10; First posted 2019-01-31 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Endothelial Dysfunction; Aging
Keywords: Polyphenols; Anthocyanins; Vascular function; Gut microbiome; Gut health; Berries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Formulation containing inert artificially colored maltodextrin, two capsules once a day, in a 500 mg capsule regimen (total intake 1000 mg)
  Interventions: Dietary Supplement: Placebo
- Aronia full spectrum - half dose (Experimental): Formulation containing 50% Aronia full spectrum and 50% placebo, two capsules once a day, in a 500 mg capsule regimen (total intake 1000 mg)
  Interventions: Dietary Supplement: Aronia full spectrum - half dose
- Aronia full spectrum - full dose (Experimental): Formulation of 100% Aronia full spectrum, two capsules once a day, in a 500 mg capsule regimen (total intake 1000 mg)
  Interventions: Dietary Supplement: Aronia full spectrum - full dose

INTERVENTIONS:
Dietary Supplement: Aronia full spectrum - half dose — Powdered whole fruit obtained from aronia berries (Aronia melanocarpa)
  Arms: Aronia full spectrum - half dose
Dietary Supplement: Aronia full spectrum - full dose — Powdered whole fruit obtained from aronia berries (Aronia melanocarpa)
  Arms: Aronia full spectrum - full dose
Dietary Supplement: Placebo — Identical formulation as the treatment consisting of colored maltodextrin using artificial colors.
  Arms: Placebo

SUMMARY:
Aging is the primary risk factor for cardiovascular disease (CVD) largely due to vascular endothelial dysfunction, a major initial step in the development of atherosclerosis. Endothelial dysfunction is characterized by impaired endothelium-dependent dilation and is primarily caused by reduced nitric oxide bioavailability secondary to oxidative stress and inflammation. Interventions that improve endothelial dysfunction are important for improving endothelial function and reducing CVD risk in this high-risk population. Aronia melanocarpa, commonly known as aronia berries or chokeberries, are rich in polyphenols such as anthocyanins, proanthocyanidins, and phenolic acids. These compounds, and derivatives resulting from gut microbial and phase II metabolism, have been shown to attenuate oxidative stress and inflammation, and to improve endothelial function. Aronia berries and other berries have been shown in numerous studies to have diverse cardiometabolic health effects including modulation of endothelial function, arterial stiffness, blood pressure, oxidative stress, and inflammation. In addition, berries, dietary fiber, polyphenols have been shown to exert positive effects on the gut microbiota, which may mediate improvements in cardiovascular health. Recently, we have demonstrated that modulation of the gut microbiota is associated with improvements in vascular dysfunction. The primary goal of the currently proposed research is to assess the efficacy and dose-dependent response of an aronia full spectrum dietary supplement to improve endothelial function in middle-aged/older men and postmenopausal women. A secondary goal is to determine whether aronia full spectrum modulation of the gut microbiota is associated with improvements in endothelial function. Other functional and biochemical measures of cardiovascular health, oxidative stress, inflammation, and polyphenol metabolism will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women (> 1 year from cessation of menstruation)
* Aged 45-75 years
* Baseline endothelial dysfunction (RHI ≤ 1.67)
* Hemoglobin A1C ≤ 6.4%
* Blood pressure < 129/80 mmHg
* Total cholesterol < 240 mg/dL
* LDL cholesterol < 190 mg/dL
* Triglycerides < 350 mg/dLhttps://register.clinicaltrials.gov/prs/app/template/Home.vm?uid=U00036MD&ts=50&sid=S0008GBU&cx=gvt3fw
* Body mass index ≥ 18.5 and < 30 kg/m2
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
* Are able to understand the nature of the study
* Able and willing to give signed written informed consent
* Signed informed consent form

Exclusion Criteria:

* Individuals taking antihypertensive, lipid-lowering, and/or hormone replacement medications
* Diagnosed hypertension, CVD, diabetes, metabolic syndrome, cancer, kidney, liver, pancreatic disease
* Obese participants, defined as BMI superior or equal to 30
* Neuropathy, thrombosis, or past arm trauma or surgery
* > 3 days/wk vigorous exercise
* Participating in a weight loss program
* Weight change > 5% in the past 3 months
* Current smokers or history of smoking in the last 12 months
* Heavy drinkers (> 7 drinks/wk for women; >14 drinks/wk for men)
* Antibiotic use at any point during the study or two months prior to enrollment
* Allergies to aronia berries or other study materials
* Unwillingness to maintain normal diet and/or physical activity pattern, or to discontinue use of dietary supplements for the duration of the study
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline reactive hyperemia index (RHI) after 6 weeks consumption | Baseline and 6 weeks
  Determine the effects on RHI measured by EndoPAT

SECONDARY OUTCOMES:
Gut microbiota analysis | Baseline and 6 weeks
  Determine the effects on stool sample microbial populations
Blood pressure | Baseline and 6 weeks
  Determine the effects on brachial and aortic blood pressure measured by SphygmoCor
Augmentation index | Baseline and 6 weeks
  Determine the effects on augmentation index measured by SphygmoCor
Gastrointestinal health | Baseline and 6 weeks
  Determine the effects on gastrointestinal health using a validated questionnaire
Pulse wave velocity | Baseline and 6 weeks
  Determine the effects on aortic arterial stiffness measured by SphygmoCor
Blood lipids | Baseline and 6 weeks
  Determine the effects on blood lipid profiles (total cholesterol, HDL, LDL, triglycerides)
Blood hemoglobin A1c | Baseline and 6 weeks
  Determine the effects on Hemoglobin A1c
Blood oxidized LDL | Baseline and 6 weeks
  Determine the effects on oxidized LDL
Blood ICAM | Baseline and 6 weeks
  Determine the effects on ICAM
Blood VCAM | Baseline and 6 weeks
  Determine the effects on VCAM

OTHER OUTCOMES:
Plasma polyphenol metabolites | Baseline and 6 weeks
  Determine the effects on plasma polyphenol metabolites
Fecal polyphenol metabolites | Baseline and 6 weeks
  Determine the effects on fecal polyphenol metabolites
Urine polyphenol metabolites | Baseline and 6 weeks
  Determine the effects on urine polyphenol metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Johnson, PhD, RDN, Principal Investigator — Department of Food Science and Human Nutrition, Colorado State University
Locations (1):
- Department of Food Science and Human Nutrition, Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No